## **COVER PAGE**

TITLE: <u>Improving Self-Efficacy</u> <u>Through a Telenovela: Feasibility Study</u>

NCT number: **NCT04533594** 

Document Date: 12/23/21

## Statistical Analysis Plan

We will describe the data to identify any patterns across the two time points (baseline and final score-up to 6 weeks). Those with and without missing data will be compared on baseline variables to determine variables related to missingness. We will group missing data reasons and run frequency distribution. We will impute any missing data. The continuous outcome measures at baseline and at final posttest assessments will be compared using a paired t-test with SPSS v24. If assumptions are reasonably met, we will run a repeated measures ANOVA. We will not have adequate power to apply more advanced methods of statistical inference; however, we will compute 95% confidence intervals (CI) for difference in means. All of these analyses together will help us in assessing feasibility and acceptability with a potential of showing efficacy on outcomes such as caregiver self-efficacy, anxiety and satisfaction. That information will be used in planning a larger fully powered randomized controlled efficacy study.

## **Reference:**

1. IBM SPSS Statistics for Windows, Version 24.0. Armonk: NYIBM corporation;. 1999.